CLINICAL TRIAL: NCT02925572
Title: Impact of Muscular Training Program on Body Composition of Overweight and Obese Teenagers: classi201c Cycling Exercise in Concentric Versus Eccentric
Brief Title: Teenagers: Impact of Eccentric eXercise Training on Overweight and Obesity
Acronym: TEXTOO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: ONAPS : Observatoire National de l'Activité Physique et de la Sédentarité (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CHU-0279; 2016-A00043-48 (Other: 2016-A00043-48)
Record Dates: First submitted 2016-09-26; First posted 2016-10-06 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Adolescents (12 to 17 Years Old); Obese (BMI>90th Percentile)
Keywords: pediatric obesity; eccentric exercise; body composition; training program
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Concentric cycling exercise (CON) (Experimental): 40 obese adolescents will be randomized into 2 groups: CON or EXC
  Interventions: Other: Cycling exercises
- eccentric cycling exercise (EXC) (Experimental): 40 obese adolescents will be randomized into 2 groups: CON or EXC
  Interventions: Other: Cycling exercises

INTERVENTIONS:
Other: Cycling exercises — All measurements are performed before and after the training program (12 weeks)

SUMMARY:
Nowadays, eccentric exercise can be realized in a dynamic way with an ergocycle which permits eccentric (ECC) lower limbs contractions at a defined power output. With this type of ergometer, O2 consumption (VO2) in ECC is three fold lower than in concentric (CON) for the same power output. Consequently, ECC program could be used in chronic disorders with limited capacities, such as obesity.

The investigators hypothesis that an eccentric training program, as it will induce higher mechanical constraints, would improve body composition, especially by reducing fat mass. This effect could be explained by an increased rest energy expenditure and a better improvement in biological parameters (particularly lipid profile and insulin-resistance) after ECC training (versus CON training).

This study aims to compare the modification of fat mass after an ECC program versus a CON program at the same VO2.. The secondary goal is to assess the physiological mechanisms involved in the modification of body composition.

DETAILED DESCRIPTION:
40 obese adolescents will be randomized into 2 groups: CON or EXC. The patients of ECC group will follow habituation sessions (2 weeks) to avoid the secondary muscular effects of high intensity eccentric exercise. The training program will last 12 weeks for the two groups. Before and after, each subjects will participate to the following measurements: total and segmental body composition (DXA), aerobic capacities (maximal incremental exercise test, VO2max), muscular lower limbs strength (isometric and isokinetic dynamometer), rest energy expenditure (indirect calorimetry), biological parameters (lipid profile, insulin-resistance), physical activity (actimetry), food intakes and quality of life (questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* Adolescent (12 to 17 years old)
* BMI>90th percentile
* Post puberty (Tanner 3 to 5)
* Inactive (<10 METS/h/week)
* No other chronic disease (cardio pulmonary, osteo articulary or muscular diseases), no surgery during the last 3 months, no genetic obesity and no contraindication to physical activity

Exclusion Criteria:

-

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
change in total body fat mass (Dual X ray Absorptiometry) | before and after the 12 weeks training program

SECONDARY OUTCOMES:
aerobic capacities (VO2max) | before and after the 12 weeks training program
isometric muscular lower limbs strength | before and after the 12 weeks training program
isokinetic muscular lower limbs strength | before and after the 12 weeks training program
rest energy expenditure (indirect calorimetry) | before and after the 12 weeks training program
biological parameters (plasma lipid profile and insulin-resistance ) | before and after the 12 weeks training program
physical activity (actimetry and questionnaires) | before and after the 12 weeks training program
food intakes (measurements and questionnaires) | before and after the 12 weeks training program
quality of life (questionnaires) | before and after the 12 weeks training program
segmental body composition (segmental fat and fat free mass, Dual X-ray Absorptiometry) | before and after the 12 weeks training program

CONTACTS AND LOCATIONS:
Overall Officials: Valérie JULIAN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Moore H, Pereira B, Fillon A, Miguet M, Masurier J, Beaulieu K, Finlayson G, Thivel D. The association between obesity severity and food reward in adolescents with obesity: a one-stage individual participant data meta-analysis. Eur J Nutr. 2024 Jun;63(4):1241-1255. doi: 10.1007/s00394-024-03348-4. Epub 2024 Feb 20. PMID 38376518
- [Derived] Julian V, Thivel D, Miguet M, Brengues C, Pereira B, Courteix D, Richard R, Duclos M. Bone response to eccentric versus concentric cycling in adolescents with obesity. Obes Res Clin Pract. 2020 Nov-Dec;14(6):554-560. doi: 10.1016/j.orcp.2020.10.002. Epub 2020 Oct 26. PMID 33121896